CLINICAL TRIAL: NCT05984654
Title: A Prospective, Open-label, Randomized, Split-ulcer Trial to Evaluate the Efficacy of Platelet-rich Plasma Therapy in the Treatment of Chronic Pyoderma Gangrenosum.
Brief Title: Autologous Platelet-Rich Plasma Therapy in the Treatment of Pyoderma Gangrenosum
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not obtain funding
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Ben H Kaffenberger, Clinical Associate Professor of Dermatology, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023H0207
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Pyoderma Gangrenosum
Keywords: platelet rich plasma; pyoderma gangrenosum
MeSH Terms: conditions — Pyoderma Gangrenosum

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Target ulcer Group 1(Injectable PRP) (Experimental): Under aseptic conditions, 2 mL of autologous PRP will be injected with 30 G needle at multiple sites in and around target ulcer approximately 1.5 cm apart at 0, 4, 8, and 12 weeks after local anesthesia.
  Interventions: Procedure: Platelet rich plasma therapy
- Target ulcer Group 2(Topical PRP) (Experimental): Under aseptic conditions, 2 mL of autologous PRP will be applied topically followed by a Platelet poor plasma solution soaked dressing on the second target ulcer at 0, 4, 8, and 12 weeks.
  Interventions: Procedure: Platelet rich plasma therapy
- Target ulcer Group 3(No treatment) (No Intervention): Target ulcer in the control group will receive standard wound care only.

INTERVENTIONS:
Procedure: Platelet rich plasma therapy — Approximately 30 ml of the patient's blood sample will be drawn from a peripheral vein in ACD (acid citrate dextrose) tubes. A double spin method will be used for the preparation of PRP.
  Note this is not a device or a medicine as this is autologous plasma.
  Arms: Target ulcer Group 1(Injectable PRP); Target ulcer Group 2(Topical PRP)

SUMMARY:
Pyoderma gangrenosum (PG) is a chronic inflammatory condition with severe painful ulcers. We hypothesize that Platelet-rich plasma(PRP) therapy derived from patient's own blood has a high concentration of endogenous growth factors, which will activate the wound-healing cascade stimulating formation of new blood vessels and collagen in PG ulcers.The goal of this study is to evaluate the efficacy and safety of autologous Platelet rich Plasma(PRP) therapy for the treatment of chronic Pyoderma Gangrenosum(PG). Researchers will also compare the efficacy of PRP therapy when used as a topical solution versus injections in and around the target ulcer/s.

DETAILED DESCRIPTION:
This is a prospective, randomized split-ulcer controlled trial that will enroll 10 adult patients with chronic pyoderma gangrenosum. In each participant, up to three separate ulcerations will be randomized into 3 comparative groups in 1:1:1 ratio to either receive monthly intralesional PRP injections or topical PRP therapy at 0, 4, 8, and 12 weeks while the third target ulcer will receive standard wound care only. In the event that only two ulcerations are present, they will be randomized to 1:1 standard care vs topical and intralesional PRP. All other ulcers, if any, will receive standard wound care during the study period. Participants will be followed up for 4 weeks after the completion of treatment period. The primary endpoint for this study will be the composite proportion of the target ulcers achieving either complete resolution or 50% reduction in the surface area at week 12.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent before participating in any study-specific activity.
2. Have a clinical diagnosis of classic PG as determined by the principal investigator based on results from clinical, histological, and laboratory assessments.
3. Have at least 2 PG ulcer characterized by 'item a' AND 3/5 features in 'item b' OR 2/5 features in 'item b' with support from one of the conditions listed in c. a. Stable or increasing size within 2 months preceding screening by patient report or documentation. b. Features such as violaceous border, undermining, cribriform scarring, pustules, peristomal location. c. Identifiable secondary systemic condition, such as IBD, arthritis, MGUS, noncancerous hematologic disease, streptococcal carriage, levamisole-tainted cocaine, Bruton's agammaglobulinemia.
4. Have at least two PG target ulcers that have an area = 2 cm2 and = 200 cm2 at screening.
5. Age at least 18 years at screening.
6. A negative pregnancy test (for females of childbearing potential) at both screening and at Day 0.
7. PARACELSUS Score for pyoderma gangrenosum of 10 or greater.

Exclusion Criteria:

1. Any condition (e.g., psychiatric illness, severe alcoholism, or drug abuse) or situation that may compromise the ability of the subject to give written informed consent, may put the subject at significant risk, may jeopardize the subject's safety after treatment, may confound the study results, or may interfere significantly with the subject's participation in the study.
2. History of malignancy within 2 years of screening other than carcinoma in situ of the cervix or adequately treated, non-metastatic, squamous, or basal cell carcinoma of the skin.
3. History of seropositivity for HIV antibody; active or carrier status of hepatitis B [surface antigen (HBsAg) positive, or core antibody (anti-HBc) positive with negative surface antibody]; active hepatitis C (i.e., not treated or not cleared spontaneously, as confirmed by HCV PCR).
4. Patients with hemodynamic instability, bleeding disorders, and/or platelet dysfunction syndrome.
5. A complete blood count will be performed for each participant at the beginning of the study and those with serum hemoglobin concentration <11 g/ dL or hematocrit <34% or platelet count<1, 00000/ml will be excluded from the study.
6. Patients with uncontrolled secondary systemic disease in the opinion of the investigator.
7. Systemic infection or active local infection requiring oral antibiotics within 2 weeks of Day 0.
8. History of the following treatments:

   1. Patients taking anticoagulant medication.
   2. Changes (addition, discontinuation, or changes in dose) in immunosuppressive medication (including cyclosporine, azathioprine, methotrexate, mycophenolate mofetil, apremilast, dapsone, or corticosteroids) and biologics (Anti-TNF or other biologic therapies) within 2 months of Day 0.
   3. Systemic corticosteroids > 20 mg per day (prednisone or prednisone equivalent) within 8 weeks of Day 0 or change in dose within 4 weeks of Day 0. Steroids may be tapered (although not increased above the Day 0 dose) during the trial as determined by the principal investigator.
   4. Intralesional corticosteroids within 8 weeks of day 0; topical immunomodulators are also not permitted.
   5. Systemic antibiotics within 2 weeks of Day 0.
   6. Hyperbaric treatment within 4 weeks of Day 0.
   7. Investigational drug or investigational device within 4 weeks of Day 0.
   8. Other treatments not described above should be maintained at a stable dose and frequency throughout the study as best as possible.
9. Major, general surgery within 3 months of screening, or anticipated general surgery during the study period.
10. Pregnancy plans to become pregnant during the study, delivery within 3 months of screening, or breastfeeding.
11. If previous use of cyclosporine or systemic corticosteroids, failure to have any stabilization/response is exclusionary. This potentially indicates the disease is not PG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of ulcers with complete healing or 50 % area reduction | 12 weeks
  Primary outcome will be the composite proportion of the target ulcers achieving either complete resolution or 50% reduction in the surface area at week 12 after treatment with either intralesional injectable or topical platelet-rich plasma therapy as compared to standard treatment

SECONDARY OUTCOMES:
Total surface area change | Week 12 and week 16
  Analysis of change in total surface area of target/total ulcers from baseline to week 12 and week 16
Patient Global Assessment (PGA) change | Week 12 and week 16
  Analysis of change Patient Global Assessment (PGA) from baseline until baseline to week 12 and week 16
Investigator Global Assessment (IGA) change | Week 12 and week 16
  Analysis of change Investigator Global Assessment (IGA) x maximum wound dimension from baseline until baseline to week 12 and week 16
Patient pain perception | Week 12 and week 16
  Analysis of change in patient pain perception using 10-point visual analog scale (VAS) from baseline to week 12 and week 16. This is a 10 point scale with higher scores indicating more severe pain.
Change in quality of life | Week 12 and week 16
  Analysis of change in patient quality of life using the dermatology life quality index (DLQI) from baseline to week 12 and week 16.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin H. Kaffenberger, MD, Principal Investigator — The Ohio State University- Dermatology
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No